CLINICAL TRIAL: NCT04282135
Title: Detection of Influenza or SARS-CoV-2 Infection by IMS of Nasal Air Sampling
Status: Completed | Type: Observational
Sponsor: Klinikum Bayreuth GmbH (Industry)
Responsible Party: Principal Investigator, Claus Steppert, Director Department of pulmonology and thoracic oncology, Klinikum Bayreuth GmbH
Other Study IDs: IMS 1
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infected: patients with detected Influenza RNA in nasopharyngeal swabs
  Interventions: Diagnostic Test: MCC IMS
- not infected: patients without detected Influenza RNA in nasopharyngeal swabs
  Interventions: Diagnostic Test: MCC IMS
- SARS CoV2: patients with SARS-Cov-2 infection
  Interventions: Diagnostic Test: MCC IMS

INTERVENTIONS:
Diagnostic Test: MCC IMS — Diagnosis by MCC IMS

SUMMARY:
Multicapillary Ion mobility spectrometry of nasal air aspirates shall be investigated as screening tool for the detection of Influenza and SARS-CoV-2- infection.

DETAILED DESCRIPTION:
Bacterial infections can be distinguished by analysis of the volatile organic compounds found in breath.

In patients with suspected Influenza infection, nasal air samples will be taken and analyzed by Multicapillary Ion mobility spectrometry (MCC IMS). Routinely all patients undergo polymerase chain reaction (PCR) analysis of nasopharyngeal swabs for Influenza.

MCC IMS spectra will be compared between infected and non infected patients by cluster analysis and discrimination analysis.

If the number of infected patients exceeds 50 an additional validation cohort will be investigated sequentially otherwise validation will be performed during the Influenza epidemic 2021.

Due to decreasing numbers of Influenza-A- Infections study was opened to also include patients with suspected SARS-CoV-2 infections.

ELIGIBILITY:
Inclusion Criteria:

* suspected Influenza infection

Exclusion Criteria:

* later than 48h after admission and detection of Influenza infection
* later than 32 days after admission and detection of SARS-CoV-2- infection
* no written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general population
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cluster Analysis of MCC IMS spectra. | immediatly after sampling
  Cluster Analysis of MCC IMS spectra will be obtained immediately after sampling

CONTACTS AND LOCATIONS:
Overall Officials: Claus Steppert, MD, Principal Investigator — Klinikum Bayreuth, Dpt. Pulmonology
Locations (1):
- Klinikum Bayreuth, Bayreuth, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steppert C, Steppert I, Sterlacci W, Bollinger T. Rapid detection of SARS-CoV-2 infection by multicapillary column coupled ion mobility spectrometry (MCC-IMS) of breath. A proof of concept study. J Breath Res. 2021 Mar 18;15(2). doi: 10.1088/1752-7163/abe5ca. PMID 33578396
- [Derived] Steppert C, Steppert I, Bollinger T, Sterlacci W. Rapid non-invasive detection of Influenza-A-infection by multicapillary column coupled ion mobility spectrometry. J Breath Res. 2020 Oct 22;15(1):011001. doi: 10.1088/1752-7163/abb762. PMID 33089824